CLINICAL TRIAL: NCT00067964
Title: Diet and Physical Activity Interactions in Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Allocation: Randomized | Purpose: Prevention
Other Study IDs: DHAIO (completed)
Record Dates: First submitted 2003-09-03; First posted 2003-09-05 (Estimated); Last update posted 2010-01-13 (Estimated); Status verified 2010-01

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Exercise; Diet

INTERVENTIONS:
Behavioral: small changes in physical activity and diet

SUMMARY:
The projects funded by this grant, primarily focus on environmental factors that promote weight-gain in the general human population, and how to modify these factors, to prevent further weight-gain in the future. In the coming years, the researchers at the University of Colorado-HSC hope to gain an understanding as to how small changes in diet and physical activity can be achieved and sustained to prevent weight-gain.

ELIGIBILITY:
* BMI: 21-26
* < 5lb. weight change in 6 mo.
* usual fat intake 25-35%
* regularly eats 3 meals/day
* no chronic health problems known to affect appetite
* either active or inactive (specific criteria do exist)
* no smoking
* women must be on bcps
* no evidence of depression, eating disorder, or restrained eater (determined from validated questionnaires).

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado-HSC Center for Human Nutrition, Denver, Colorado, United States